CLINICAL TRIAL: NCT04279782
Title: Investigation on Clinical Features of Suspected and Confirmed Patients of 2019 Novel Coronavirus Infection in Isolation Unit
Brief Title: Clinical Features of Suspected and Confirmed Patients of 2019 Novel Coronavirus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: XWX3
Record Dates: First submitted 2020-02-15; First posted 2020-02-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Coronavirus
Keywords: 2019 Novel Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exclusion group: Patients with two consecutive negative results of detection for 2019 Novel Coronavirus nucleic acid from pharyngeal swabs
  Interventions: Other: Comprehensive treatment
- Confirmed group: Patients with positive result of detection for 2019 Novel Coronavirus nucleic acid from pharyngeal swab
  Interventions: Other: Comprehensive treatment

INTERVENTIONS:
Other: Comprehensive treatment — Comprehensive treatment includes antiviral therapy, antibiotics therapy, symptomatic treatment, supportive therapy.

SUMMARY:
Outbreak of 2019 Novel Coronavirus infection started in Wuhan and quickly spread to the world. Suspected patients were isolated and treated in our department. Clinical data was recorded to investigate the clinical features of patients confirmed and excluded diagnosed of 2019 Novel Coronavirus infection.

DETAILED DESCRIPTION:
Medical date of suspected patients of 2019 Novel Coronavirus infection, who came to outpatient department of the Third Affiliated Hospital of Sun Yat-sen University, were sent to an expert group if they met the inclusion criteria. The expert group discussed and made a decision if the patient would be admission to isolation unit. Pharyngeal swabs of the patients were obtained and sent to local Center for Disease Control and Prevention (CDC) for detection the 2019 Novel Coronavirus after patients were admission to isolation unit. Diagnosis of 2019 Novel Coronavirus infection was confirmed if the result was positive or excluded if two consecutive results were negative. Patients' demographic data and clinical characteristics were recorded. Clinical characteristics including epidemiological history, past history, personal history, symptoms, signs, blood cells count, biochemical test results, chest computed tomography (CT) images and treatment. Comprehensive treatments were given to the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Epidemiological history including resident of Hubei province, or travel history to Hubei province or exposure to suspected patients in the past two weeks.
2. Symptoms like fever, fatigue, myalgia, headache, cough, sputum production, chest tightness, dyspnea, etc.
3. White blood cells decreased or were normal, or lymphocytes decreased, and chest CT images showed typical findings of viral pneumonia.

Exclusion Criteria:

1. Patients can not follow-up;
2. Investigator considering inappropriate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Suspected patients of 2019 Novel Coronavirus infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 28 days
  If the patient will survive after comprehensive treatment

SECONDARY OUTCOMES:
Chest computed tomography | 28 days
  Images of chest computed tomography are obtained to find out the changes in the course of treatment
Recovery Time | 28 days
  Time for recovery from admission to discharged
Depression evaluation | 28 days
  A self-rating depression scale (SCL-90) will be finished from patients and medical staff. There are 90 questions. Each question scores from 1 to 5. Minimum score is 90, maximun score is 450. High scores indicate poor condition.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng L, Liu J, Xu W, Luo Q, Chen D, Lei Z, Huang Z, Li X, Deng K, Lin B, Gao Z. SARS-CoV-2 can be detected in urine, blood, anal swabs, and oropharyngeal swabs specimens. J Med Virol. 2020 Sep;92(9):1676-1680. doi: 10.1002/jmv.25936. Epub 2020 Apr 30. PMID 32330305